CLINICAL TRIAL: NCT06772246
Title: A Single Blind, Fixed Sequence, Single-dose Study to Evaluate the Serious Risk of QTc Prolongation With Quizartinib in Healthy Subjects Under Rapid Acceleration of Heart Rate
Brief Title: A Study to Evaluate QTc Prolongation With Quizartinib in Healthy Subjects Under Rapid Acceleration of Heart Rate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC220-165
Record Dates: First submitted 2024-12-13; First posted 2025-01-13 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Healthy Subjects
Keywords: quizartinib
MeSH Terms: interventions — quizartinib

STUDY DESIGN:
Masking Description: This is a single-blinded study where only the participants will be blinded to the treatment being administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Healthy Participants (Experimental): All participants will receive either an oral dose of 90 mg of quizartinib or placebo on Day 1. On Day 2, all participants will receive the treatment that was not given on Day 1.
  Interventions: Drug: Quizartinib; Other: Placebo

INTERVENTIONS:
Drug: Quizartinib — Participants will receive a single oral dose of 90 mg
  Other Names: VANFLYTA®
Other: Placebo — Participants will receive a single oral dose of 90 mg

SUMMARY:
This study will evaluate the impact of rapid acceleration in the heart rate on the QT prolongation of quizartinib.

DETAILED DESCRIPTION:
This is a QT assessment study of quizartinib when given as a single oral dose of 90 mg in 70 healthy subjects.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male and female subjects 18 to 55 years of age (inclusive), with a BMI of 18 kg/m2 to 32 kg/m2 (inclusive) with a minimum body weight of 40 kg at Screening.
2. Has vital signs (measured after subject has been supine for at least 5 minutes) at Screening within the following ranges: heart rate: 50-100 beats per minute (bpm); systolic blood pressure (BP): 90-145 mmHg; diastolic BP: 50-95 mmHg. Out-of-range vital signs may be repeated once.
3. Liver function test results (alanine aminotransferase [ALT], aspartate aminotransferase [AST], and total bilirubin [TBil]) must be equal to or below the upper limit of normal.
4. Hemoglobin levels must ≥11.5 g/dL for female subjects and ≥12.5 g/dL for male subjects.
5. In females, documented surgical sterilization (ie, documented hysterectomy, bilateral tubal ligation, or bilateral salpingo-oophorectomy, Essure® with hysterosalpingogram [documentation to confirm tubal occlusion 12 weeks after procedure]), postmenopausal status for at least 1 year (follicle stimulating hormone [FSH] > 40 mIU/mL serum and estradiol <40 pg/mL [<147 pmol/L] at Screening), or agreement to have a sterile male partner, or agreement to use 1 of the protocol-approved means of contraception from Screening until 7 months after the dose of quizartinib.
6. In males, documented surgical sterilization, or sexual abstinence, or agreement to use 1 of the protocol-approved means of contraception from Screening until 4 months after the single dose of quizartinib.

Key Exclusion Criteria:

1. Any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormality) that could interfere with subject's safety, obtaining informed consent, compliance to the study procedures, or the validity of the study results.
2. In the opinion of the investigator, history of a clinically significant illness within 4 weeks prior to administration of quizartinib.
3. History or presence of an abnormal ECG, which, in the investigator's opinion, is clinically significant and/or a QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 milliseconds (ms) at Screening
4. Females who are pregnant or breastfeeding
5. Laboratory results (serum chemistry, hematology, and urinalysis) outside the normal range, if considered clinically significant by the investigator. Estimated creatinine clearance (CrCl) < 90 mL/min (calculated by Cockcroft-Gault equation) at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2024-10-24 (Actual); Primary Completion 2025-06-12 (Actual); Study Completion 2025-06-12 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate | Day 1 and Day 2

SECONDARY OUTCOMES:
Treatment Emergent Adverse Events (TEAEs) | From Day 1 up to the last day of Safety Follow-up (approximately 16 days)
  TEAEs are defined as new AEs that occur after the first dose of study drug, including 14 days after last dose of study drug" to end of the sentence
Pharmacokinetic Parameter: Cmax | Days 1, 2 and 3
  Maximum concentration, determined directly from individual concentration-time data
Pharmacokinetic Parameter: Tmax | Days 1, 2 and 3
  Time of the maximum concentration
Pharmacokinetic Parameter: AUClast | Days 1, 2 and 3
  Area under the concentration-time curve from time-zero to the time of the last quantifiable concentration; calculated using the linear up log down

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (1):
- WCT, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No